CLINICAL TRIAL: NCT05847127
Title: Is There a Difference in Pulmonary Functions and Craniovertebral Angle Among Adolescent Based on Their Smart Phone Usage Time? A Cross Sectional Study
Brief Title: Is There a Difference in Pulmonary Functions and Craniovertebral Angle Among Adolescent Based on Smart Phone Usage
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maryan Mamdouh Fayez (Other)
Responsible Party: Sponsor-Investigator, Maryan Mamdouh Fayez, Lecturer at Department of Physical Therapy for Pediatrics, Egyptian Chinese University
Organization: Egyptian Chinese University (Other)
Other Study IDs: P.T.REC/012/003908
Record Dates: First submitted 2023-02-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Function Tests
Keywords: Pulmonary function; craniovertebral angle; smart phone usage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The smartphones have become a necessity for most adolescents as they are used for communication and entertainment and education purposes especially in the period of COVID pandemic. They spend most of their time in using smartphones. This could have side effects on their health.

While using a smartphone, adolescent usually flex their neck and maintain the head in a forward position for long periods of time, which may affect the craniovertebral angle and pulmonary functions as sustained forward neck posture may lead to respiratory dysfunction.The purpose of the study is to investigate the effect of smart phones and tablets usage time on craniovertebral angle and problems of pulmonary functions among adolescents between 14-18 years' old.

DETAILED DESCRIPTION:
A well-developed adolescents of both genders will participate in this study after signing institutionally approved consent form prior to data collection

* They will be recruited from many secondary schools in Cairo. Their ages range from 14 to 18 years. They will be subdivided into two groups according to Smartphone addiction scale-short version (SAS-SV) into an addict group who use smart phone not less than 4 hours/day for at least 4 years and non-addict group who used smart phone less than that.
* Design of the study: Cross sectional design will be applied in this study.
* Smartphone addiction scale-short version (SAS-SV) will be used to divide the subjects into two groups addict and non-addict groups
* (Image J) image processing and analysis in Java system will be used to measure the craniovertebral angle for both groups.
* Micromedical Gold standard fully computerized portable auto spirometer will be used to measure Pulmonary functions test in the form of forced expiratory volume in one second (FEV1), forced vital capacity (FVC)and FEV1/FVC for both groups.
* All data will be recorded and statistically analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of late childhood ( adolescence)
* Age of participants ranged from 14 to 18 years.
* Subjects with normal development.

Exclusion Criteria:

* Athletic one.
* Genetic spinal deformity.
* Injury to the neck.
* History of inflammatory joint disease.
* History of surgical intervention at the neck. Patients with neuropediatric problem.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Well-developed adolescents of both genders.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function tests | Baseline
  FVC & FEV1 both are measured in liters
Craniovertebral angle | Baseline
  measured in degree
Pulmonary function tests | Baseline
  FEV1/FVC measured in percentage ( % )

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian Chinese University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided